CLINICAL TRIAL: NCT04306302
Title: A Randomized, Double-blind, Phase 1 Study to Evaluate the Safety, Reactogenicity, and Immunogenicity of Different Doses of VAC52416 (ExPEC10V) in Japanese Adults Aged 60 to 85 Years
Brief Title: A Study to Evaluate the Different Doses of VAC52416 (ExPEC10V) in Japanese Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: CR108778; VAC52416BAC1002 (Other: Janssen Pharmaceutical K.K.)
Record Dates: First submitted 2020-03-11; First posted 2020-03-12 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medium-dose ExPEC10V or Placebo: Group 1 (Experimental): Participants will be randomized to receive a single intramuscular (IM) injection of medium dose of ExPEC10V or Placebo on Day 1.
  Interventions: Biological: ExPEC10V; Biological: Placebo
- High-dose ExPEC10V or Placebo: Group 2 (Experimental): Participants will be randomized to receive a single IM injection of high dose (based on safety assessment through Day 15 postvaccination of medium dose) of ExPEC10V or Placebo on Day 1.
  Interventions: Biological: ExPEC10V; Biological: Placebo

INTERVENTIONS:
Biological: ExPEC10V — Participants will receive a single IM injection of ExPEC10V.
  Other Names: VAC52416
Biological: Placebo — Participants will receive single IM injection of matching placebo.

SUMMARY:
The purpose of this study is to evaluate the safety and reactogenicity of different doses of extraintestinal pathogenic Escherichia coli 10 valent (ExPEC10V) in Japanese participants greater than or equal to (>=) 60 to less than or equal to (<=) 85 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be Japanese as determined by participant's verbal report
* Must be healthy or medically stable, in the investigator's clinical judgment, as confirmed by medical history, physical examination, vital signs, 12-lead electrocardiogram (ECG), and clinical laboratory tests performed at the screening visit
* Willing and able to adhere to the lifestyle restrictions
* Agrees not to donate blood until 12 weeks after receiving the study intervention
* Must be willing to provide verifiable identification, has means to be contacted, and to contact the investigator during the study

Exclusion Criteria:

* Clinically significant illness (this does not include minor illnesses such as diarrhea or mild upper respiratory tract infection) or temperature greater than or equal to (>=) 38.0 degree Celsius (100.4 degree Fahrenheit ) within 24 hours prior to the administration of study intervention; enrollment at a later date is permitted (provided the screening window of 28 days is respected)
* History of malignancy within 5 years before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy, which is considered cured with minimal risk of recurrence)
* Known allergies, hypersensitivity, or intolerance to ExPEC10V or its excipients
* Known allergy or history of anaphylaxis or other serious adverse reactions to vaccines or vaccine excipients
* Contraindication to Intramuscular (IM) injections and blood draws example, bleeding disorders

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-03-13 (Actual); Primary Completion 2020-12-24 (Actual); Study Completion 2020-12-24 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Solicited Local Adverse Events (AEs) Collected for 14 days post-Vaccination | 14 days post-Vaccination (Up to Day 15)
  Number of participants with solicited local AEs will be reported. Solicited local AEs (pain/tenderness, erythema, and swelling at the injection site) and will be noted in the participant diary for 14 days post-vaccination.
Number of Participants with Solicited Systemic AEs Collected for 14 days post-Vaccination | 14 days post-Vaccination (Up to Day 15)
  Number of participants with solicited systemic AEs will be reported. Solicited systemic AEs (oral body temperature, headache, fatigue, nausea, and myalgia) will be noted in the participant diary for 14 days post-vaccination.
Number of Participants with Unsolicited AEs From the Administration of Study Vaccine until 29 Days post-Vaccination | From the administration of study vaccine until 29 days post-Vaccination (Up to Day 30)
  Number of participants with unsolicited AEs will be reported. Unsolicited AEs are all AEs for which the participant is not specifically questioned in the participants diary.
Number of Participants with Serious AEs from the Administration of the Study Vaccine until Day 181 | From the administration of study vaccine until 180 days post-Vaccination (Up to Day 181)
  Number of participants with SAEs will be reported. A SAE is any AE that results in: death, persistent or significant disability/incapacity, requires inpatient hospitalization or prolongation of existing hospitalization, is life threatening experience, is a congenital anomaly/birth defect, is suspected transmission of any infectious agent via a medicinal product, is medically important, and may jeopardize participant or may require medical or surgical intervention to prevent one of the outcomes listed above.

SECONDARY OUTCOMES:
Antibody Titers for ExPEC10V as Determined by Multiplex ECL-based Immunoassay | Days 15 and 30
  Antibody titers for ExPEC10V will be determined by multiplex ECL-based immunoassay.
Antibody Titers for ExPEC10V as Determined by Multiplex Opsonophagocytic Assay (MOPA) | Day 15 and 30
  Antibody titers for ExPEC10V will be determined by MOPA.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (1):
- SOUSEIKAI PS Clinic, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency